CLINICAL TRIAL: NCT06411093
Title: A Single-center, Randomized, Open-labelled Trial to Evaluate the Efficacy and Safety of the Kinesiology Tape for the Treatment of Paronychia Induced by Epidermal Growth Factor Receptor Inhibitors in Cancer Patients
Brief Title: Efficacy and Safety of Kinesiology Tape Wrapping for Paronychia Induced by Epidermal Growth Factor Receptor Inhibitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202001747A3
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Paronychia; Epidermal Growth Factor Receptor Inhibitor
MeSH Terms: conditions — Paronychia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A combination of Kinesiology tape wrapping and conventional treatment (Experimental): Patients in the intervention arm will receive Kinesiology tape wrapping to separate the nail plate from the inflamed periungual tissue in addition to conventional treatment. This intervention will be applied at outpatient visits or during hospitalization. If the Kinesiology tape falls off, patients can either replace it themselves or leave it off until the next outpatient visit or unexpected hospitalization.
  Interventions: Combination Product: Kinesiology tape wrapping; Drug: Conventional treatment including silver nitrate cauterization
- Conventional treatment (Active Comparator): Patients in this arm will receive management according to routine clinical practice, including chemical cauterization with silver nitrate, with or without topical antiseptics, topical steroids, topical beta-blockers, systemic steroids, and systemic antibiotics. The above treatment will be applied at outpatient visits or during hospitalization.
  Interventions: Drug: Conventional treatment including silver nitrate cauterization

INTERVENTIONS:
Combination Product: Kinesiology tape wrapping — Place Kinesiology tape between the nail plate and the inflamed periungual granulation tissue in addition to conventional treatment for 3 months
  Other Names: "NITTO"Medical Adhesive Tape (Non-Sterile)
  Arms: A combination of Kinesiology tape wrapping and conventional treatment
Drug: Conventional treatment including silver nitrate cauterization — Conventional treatment including silver nitrate cauterization, with or without topical antiseptics, topical steroids, topical beta-blockers, short-term systemic antibiotics, systemic steroids for 3 months

SUMMARY:
Epidermal growth factor receptor inhibitors(EGFRIs) have been applied in several common malignancies including advanced non-small cell lung cancer. Paronychia is one of the most common cutaneous side effects, characterized by inflamed granulation tissue around the nails leading to pain and reduced quality of life. Despite available conventional therapies such as topical beta-blockers or chemical cauterization, some patients still do not respond well. Our previous pilot study suggested that adding Kinesiology tape wrapping to the conventional treatment may effectively improve pain and granulomas in patients with treatment-resistant EGFRI-related paronychia, with good safety. This study aims to evaluate the clinical efficacy and safety of using Kinesiology tape wrapping as an adjunct to conventional therapy for patients with EGFRI-related paronychia.

DETAILED DESCRIPTION:
In this study, eligible patients with paronychia affecting their big toes will be included and randomized to receive a combination of Kinesiology tape wrapping and conventional treatment, or conventional treatment alone for 3 months. Patients are evaluated at baseline, at 1, 2, 4, 8, and 12 weeks after the initiation of the treatment. These evaluations will occur at the outpatient department or through phone contact and photos taken by patients if they cannot visit in person. Efficacy endpoints include pain numerical rating scale (NRS) and scoring system for paronychia related to oncologic treatments (SPOT). Besides, any side effects will be recorded at each visit.

ELIGIBILITY:
Inclusion Criteria:

* EGFR inhibitors-induced paronychia
* Having at least one big toe involved with CTCAE(Common Terminology Criteria for Adverse Events) grade 2-3 paronychia

Exclusion Criteria:

* Younger than 20 years
* severe ingrown nails
* concomitant cutaneous infection
* severe nail destruction
* chronic paronychia with severe periungual fibrosis

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the severity of pain by Numerical Rating Scale | Evaluated at week 1, 2, 4, 6, 8 and 12 after the initiation of intervention
  Patients rate the severity of pain over the tender point of the affected big toe on a scale of 0 to 10, with 0 being no pain at all and 10 being the worst pain imaginable.
Change in the severity of paronychia by the scoring system for paronychia related to oncologic treatments (SPOT) | Evaluated at week 2, 4, 6, 8 and 12 after the initiation of intervention
  The SPOT evaluates the severity of the affected big toe based on four parameters, including redness, edema, discharge and granulation tissue, each measured on a 4-point scale from 0 to 3 with 0 for no presence of signs and 3 for most severe of lesions. The total score ranges from 0 to 12.

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Jung Hsu, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Hsu TJ, Yeh HH, Liu KL. Kinesiology tapes wrapping for paronychia induced by epidermal growth factor receptor inhibitors: A pilot study. Dermatol Ther. 2022 Jun;35(6):e15463. doi: 10.1111/dth.15463. Epub 2022 Mar 29. No abstract available. PMID 35307912